CLINICAL TRIAL: NCT04970979
Title: Influencing Factors of Exercise Adherence in Home-based Cardiac Rehabilitation in Patients With Coronary Artery Disease
Brief Title: Exercise Adherence in Home-based Cardiac Rehabilitation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006761-M2021057
Record Dates: First submitted 2021-06-27; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-06

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Home-based cardiac rehabilitation; Exercise adherence
MeSH Terms: conditions — Coronary Artery Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with coronary artery disease: patients with coronary artery disease
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — questionnaire about the influencing factors of home-based cardiac rehabilitation

SUMMARY:
The study will investigate the influencing factors of exercise adherence of home-based cardiac rehabilitation in patients with coronary artery disease.

DETAILED DESCRIPTION:
The study will conduct a quantitative questionnaire survey. Patients with coronary artery disease in home-based cardiac rehabilitation will receive investigation of the influencing factors of exercise adherence.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of coronary artery disease;
* Age ≤75 years old;
* Participated in home-based cardiac rehabilitation ≥12 weeks;
* Volunteer to participate in this study.

Exclusion Criteria:

* Have other serious acute or chronic diseases;
* Have severe audio-visual or speech impairments that may affect understanding and answering questions.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-07-18 (Estimated); Primary Completion 2022-02-18 (Estimated); Study Completion 2022-02-18 (Estimated)

PRIMARY OUTCOMES:
Influencing factors of exercise adherence | The influencing factors of exercise adherence in home-based cardiac rehabilitation will be measured by the Theory of Planned Behavior Questionnaire through study completion, an average of 1 year
  Influencing factors of exercise adherence in home-based cardiac rehabilitation
Exercise adherence | The exercise adherence will be measured by the Home-based Exercise Training Adherence Questionnaire through study completion, an average of 1 year
  Adherence of home-based exercise training

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided